CLINICAL TRIAL: NCT06141603
Title: Comparison of Upper and Lower Limb Maximal Exercise Capacities, Muscle Oxygenation and Energy Consumption During Tests in Patients With Interstitial Lung Disease
Brief Title: Comparison of Upper and Lower Limb Maximal Exercise Capacities and Muscle Oxygenation in Patients With ILD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Study director, PT, PhD, Prof.Dr. Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Head of Cardiopulmonary Rehabilitation Clinic, Gazi University
Other Study IDs: Gazi University 28
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Interstitial Lung Disease
Keywords: interstitial lung disease; muscle oxygenation; cardiopulmonary exercise testing
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lower Extremity Group: The first test is the cardiopulmonary exercise test (CPET), which evaluates the maximal exercise capacity of the lower extremities and will be performed on a treadmill.
  During the test, the muscle oxygen of the individuals will be measured with a near-infrared spectrometer, and their energy consumption will be measured with a multisensory physical activity monitor.
- Upper Extremity Group: In the second test, the maximal exercise capacity for the upper limb will again be evaluated by CPET and performed on the arm ergometer.
  The second test will be conducted 48 hours after the lower extremity exercise test.
  During the test in the second group, as in the first test, muscle oxygen will be measured with a near-infrared spectrometer, and energy expenditure with a multisensory physical activity monitor.

SUMMARY:
Interstitial lung diseases (ILD) are a complex group of diseases that cause significant morbidity and mortality, develop diffuse lung parenchyma and alveolar inflammation, as well as interstitial fibrosis, which refers to more than 200 diseases. Due to restrictive type ventilation disorder and impaired pulmonary gas exchange, pulmonary function has deteriorated in these patients and progressive shortness of breath, fatigue, cough and exercise intolerance are usually observed, which also affects the quality of life.

DETAILED DESCRIPTION:
As a result of the chronic inflammatory process of the disease, structural and mechanical pulmonary disorders develop, which are cited as the causes of deterioration in cardiopulmonary functions. In these patients, there is a decrease in static and dynamic lung volumes and carbon monoxide diffusion capacity. As a result of this mechanism, the level of physical activity decreases due to increased shortness of breath during activity. In ILD, there is a decrease in peripheral November muscle strength of both the upper extremities and lower extremities. November it was stated that the weakness of the skeletal muscles of the lower extremities was more pronounced than the skeletal muscles of the upper extremities due to disuse in these patients, and the muscle strength of the upper extremities did not decrease significantly. However, it has been reported that upper limb exercise capacity is worse than lower limb exercise capacity. Arterial hypoxemia is shown as the main reason for the decrease in exercise performance, and peak oxygen consumption (VO2peak) decreased in these patients.

In healthy people, respiratory frequency, tidal volume (VT), minute ventilation and oxygen consumption increase during exercise. In interstitial lung patients, vital capacity decreases at rest, which leads to limitation of VT. Lung compliance decreases and respiratory workload increases. The respiratory workload, which increases even more during exercise, has a bad effect on ventricular function. This causes a lower oxygen pulse and pulse volume in patients during exercise than in healthy individuals.

The primary aim of the study: To compare the maximal exercise capacities and muscle oxygenation during cardiopulmonary exercise tests of upper and lower extremities in patients with interstitial lung disease.

The secondary aim of the study is to compare energy consumption and the perception of dyspnea and fatigue during tests in patients with interstitial lung disease.

The primary outcome will be upper and lower maximal exercise capacities (cardiopulmonary exercise tests) and muscle oxygenation during cardiopulmonary exercise tests (Near-infrared spectroscopy) device).

Secondary outcome will be energy consumption (multi sensor activity device), the perception of dyspnea (Modified Borg Scale (MBS)) and fatigue (MBS).

ELIGIBILITY:
Inclusion Criteria:

* patients between the ages of 18-75 with interstitial lung disease

Exclusion Criteria:

* acute infection during the study
* have an orthopedic or neurological disease that will affect their exercise capacity
* acute exacerbation or any infection
* have contraindications to the exercise test
* an acute respiratory infection
* had Coronavirus-19 (COVID-19) disease in the last 3 months
* have undergone different treatments other than standard medical treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients diagnosed with interstitial lung disease will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Peripheral Muscle Oxygenation | through study completion, an average of 1 year
  Peripheral muscle oxygen will be measured by near-infrared spectrometry. The device probes will be placed on the upper and lower extremities for both tests.
  The device allows to display of the percentage of oxygen, the concentration of oxyhemoglobin, and deoxyhemoglobin, the difference between oxyhemoglobin and deoxyhemoglobin, and the total hemoglobin. These parameters will be evaluated in our study.

SECONDARY OUTCOMES:
Maximal Exercise Capacity | through study completion, an average of 1 year
  Maximal Exercise capacity will be evaluated with Cardiopulmonary Exercise testing. The Cardiopulmonary Exercise Testing will be applied according to American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Energy Consumption During Tests | through study completion, an average of 1 year
  Energy consumption will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wear the multi sensor physical activity monitor over the triceps muscle of the non-dominant arm during CPETs. Energy consumption (joule / day) will be measured with the multi-sensor physical activity monitor. The measured parameter will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical Activity Level (Total energy expenditure) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Total energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Active energy expenditure (joule / day)) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Active energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Physical activity time (min / day)) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Physical activity time (min / day)will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Average metabolic equivalent (MET / day)) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Average metabolic equivalent (MET / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Number of steps (steps / day)) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Number of steps (steps / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Time spent lying down (min / day) days)) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Time spent lying down (min / day) days) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Sleep time (min / day)) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Sleep time (min / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Peripheral Muscle Strength | through study completion, an average of 1 year
  Isometric peripheral muscle strength will be measured with a portable hand dynamometer (JTECH Commander, USA).
  Measurements will be repeated on the shoulder abductors and knee extensors three times on the right and left.
Dyspnea | through study completion, an average of 1 year
  Modified Borg Scale: The Modified Borg scale is a subjective scale that scores 0-10 for breathlessness and fatigue at rest and/or during activity. The lowest 0 points "not at all" the highest 10 points "very severe" means shortness of breath.
Fatigue | through study completion, an average of 1 year
  Fatigue will be measured by the Turkish adaptation of the Fatigue Severity Scale. The Fatigue Severity Scale (FSS) is a scale that evaluates fatigue and consists of 9 questions. Scores can be taken from the scale in the range of 0 to 63 points. Each item is scored between 0 and 7 points. The total score is divided by 9 and if the average is less than 4, there is no fatigue, and if more than 4 points, it is considered that there is fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Beyza Nur ÖYMEZ, Pt., Principal Investigator — Gazi University; Nilgün YILMAZ DEMİRCİ, Prof. Dr., Principal Investigator — Gazi University; Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guler SA, Corte TJ. Interstitial Lung Disease in 2020: A History of Progress. Clin Chest Med. 2021 Jun;42(2):229-239. doi: 10.1016/j.ccm.2021.03.001. PMID 34024399
- [Background] Mikolasch TA, Garthwaite HS, Porter JC. Update in diagnosis and management of interstitial lung disease . Clin Med (Lond). 2017 Apr;17(2):146-153. doi: 10.7861/clinmedicine.17-2-146. PMID 28365626
- [Background] Molgat-Seon Y, Schaeffer MR, Ryerson CJ, Guenette JA. Exercise Pathophysiology in Interstitial Lung Disease. Clin Chest Med. 2019 Jun;40(2):405-420. doi: 10.1016/j.ccm.2019.02.011. PMID 31078218
- [Background] Bourke SJ. Interstitial lung disease: progress and problems. Postgrad Med J. 2006 Aug;82(970):494-9. doi: 10.1136/pgmj.2006.046417. PMID 16891438
- [Background] Shen Q, Guo T, Song M, Guo W, Zhang Y, Duan W, Peng Y, Ni S, Ouyang X, Peng H. Pain is a common problem in patients with ILD. Respir Res. 2020 Nov 11;21(1):297. doi: 10.1186/s12931-020-01564-0. PMID 33176795
- [Background] Tomlinson OW, Markham L, Wollerton RL, Knight BA, Duckworth A, Gibbons MA, Scotton CJ, Williams CA. Validity and repeatability of cardiopulmonary exercise testing in interstitial lung disease. BMC Pulm Med. 2022 Dec 22;22(1):485. doi: 10.1186/s12890-022-02289-0. PMID 36550475
- [Background] Dowman LM, McDonald CF, Hill CJ, Lee AL, Barker K, Boote C, Glaspole I, Goh NSL, Southcott AM, Burge AT, Gillies R, Martin A, Holland AE. The evidence of benefits of exercise training in interstitial lung disease: a randomised controlled trial. Thorax. 2017 Jul;72(7):610-619. doi: 10.1136/thoraxjnl-2016-208638. Epub 2017 Feb 17. PMID 28213592
- [Background] Antoniou KM, Margaritopoulos GA, Tomassetti S, Bonella F, Costabel U, Poletti V. Interstitial lung disease. Eur Respir Rev. 2014 Mar 1;23(131):40-54. doi: 10.1183/09059180.00009113. PMID 24591661
- [Background] Baydur A. Pulmonary physiology in interstitial lung disease: recent developments in diagnostic and prognostic implications. Curr Opin Pulm Med. 1996 Sep;2(5):370-5. doi: 10.1097/00063198-199609000-00005. PMID 9363170
- [Background] Panagiotou M, Church AC, Johnson MK, Peacock AJ. Pulmonary vascular and cardiac impairment in interstitial lung disease. Eur Respir Rev. 2017 Jan 17;26(143):160053. doi: 10.1183/16000617.0053-2016. Print 2017 Jan. PMID 28096284
- [Background] Nishiyama O, Yamazaki R, Sano H, Iwanaga T, Higashimoto Y, Kume H, Tohda Y. Physical activity in daily life in patients with idiopathic pulmonary fibrosis. Respir Investig. 2018 Jan;56(1):57-63. doi: 10.1016/j.resinv.2017.09.004. Epub 2017 Oct 23. PMID 29325683
- [Background] Mendes P, Wickerson L, Helm D, Janaudis-Ferreira T, Brooks D, Singer LG, Mathur S. Skeletal muscle atrophy in advanced interstitial lung disease. Respirology. 2015 Aug;20(6):953-9. doi: 10.1111/resp.12571. Epub 2015 Jun 17. PMID 26081374
- [Background] Harris-Eze AO, Sridhar G, Clemens RE, Zintel TA, Gallagher CG, Marciniuk DD. Role of hypoxemia and pulmonary mechanics in exercise limitation in interstitial lung disease. Am J Respir Crit Care Med. 1996 Oct;154(4 Pt 1):994-1001. doi: 10.1164/ajrccm.154.4.8887597.
- [Background] Bhambhani Y, Maikala R, Buckley S. Muscle oxygenation during incremental arm and leg exercise in men and women. Eur J Appl Physiol Occup Physiol. 1998 Oct;78(5):422-31. doi: 10.1007/s004210050441. PMID 9809843
- [Background] Molgat-Seon Y, Schaeffer MR, Ryerson CJ, Guenette JA. Cardiopulmonary Exercise Testing in Patients With Interstitial Lung Disease. Front Physiol. 2020 Jul 10;11:832. doi: 10.3389/fphys.2020.00832. eCollection 2020. PMID 32754054
- [Background] Orr JL, Williamson P, Anderson W, Ross R, McCafferty S, Fettes P. Cardiopulmonary exercise testing: arm crank vs cycle ergometry. Anaesthesia. 2013 May;68(5):497-501. doi: 10.1111/anae.12195. PMID 23573845
- [Background] Franssen FM, Wouters EF, Baarends EM, Akkermans MA, Schols AM. Arm mechanical efficiency and arm exercise capacity are relatively preserved in chronic obstructive pulmonary disease. Med Sci Sports Exerc. 2002 Oct;34(10):1570-6. doi: 10.1097/00005768-200210000-00007. PMID 12370557
- [Background] Lollgen H, Leyk D. Exercise Testing in Sports Medicine. Dtsch Arztebl Int. 2018 Jun 15;115(24):409-416. doi: 10.3238/arztebl.2018.0409. PMID 29968559
- [Background] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Background] Johnson JD, Theurer WM. A stepwise approach to the interpretation of pulmonary function tests. Am Fam Physician. 2014 Mar 1;89(5):359-66. PMID 24695507
- [Background] Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung volumes and forced ventilatory flows. Eur Respir J. 1993 Mar;6 Suppl 16:5-40. doi: 10.1183/09041950.005s1693. No abstract available. PMID 24576915
- [Background] Subudhi AW, Dimmen AC, Roach RC. Effects of acute hypoxia on cerebral and muscle oxygenation during incremental exercise. J Appl Physiol (1985). 2007 Jul;103(1):177-83. doi: 10.1152/japplphysiol.01460.2006. Epub 2007 Apr 12. PMID 17431082
- [Background] Lusina SJ, Warburton DE, Hatfield NG, Sheel AW. Muscle deoxygenation of upper-limb muscles during progressive arm-cranking exercise. Appl Physiol Nutr Metab. 2008 Apr;33(2):231-8. doi: 10.1139/h07-156. PMID 18347677
- [Background] Lee JA, Laurson KR. Validity of the SenseWear armband step count measure during controlled and free-living conditions. J Exerc Sci Fit. 2015 Jun;13(1):16-23. doi: 10.1016/j.jesf.2014.11.002. Epub 2015 Jan 29. PMID 29541094
- [Background] Patel SA, Benzo RP, Slivka WA, Sciurba FC. Activity monitoring and energy expenditure in COPD patients: a validation study. COPD. 2007 Jun;4(2):107-12. doi: 10.1080/15412550701246658. PMID 17530503
- [Background] Ross RM. ATS/ACCP statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 May 15;167(10):1451; author reply 1451. doi: 10.1164/ajrccm.167.10.950. No abstract available. PMID 12738602
- [Background] Pane C, Salzano A, Trinchillo A, Del Prete C, Casali C, Marcotulli C, Defazio G, Guardasole V, Vastarella R, Giallauria F, Puorro G, Marsili A, De Michele G, Filla A, Cittadini A, Sacca F. Safety and feasibility of upper limb cardiopulmonary exercise test in Friedreich ataxia. Eur J Prev Cardiol. 2022 Mar 25;29(3):445-451. doi: 10.1093/eurjpc/zwaa134. PMID 33624001
- [Background] Andrews AW, Thomas MW, Bohannon RW. Normative values for isometric muscle force measurements obtained with hand-held dynamometers. Phys Ther. 1996 Mar;76(3):248-59. doi: 10.1093/ptj/76.3.248. PMID 8602410
- [Background] Bohannon RW. Reference values for extremity muscle strength obtained by hand-held dynamometry from adults aged 20 to 79 years. Arch Phys Med Rehabil. 1997 Jan;78(1):26-32. doi: 10.1016/s0003-9993(97)90005-8. PMID 9014953
- [Background] Wilson RC, Jones PW. A comparison of the visual analogue scale and modified Borg scale for the measurement of dyspnoea during exercise. Clin Sci (Lond). 1989 Mar;76(3):277-82. doi: 10.1042/cs0760277. PMID 2924519
- [Background] Mahler DA, Rosiello RA, Harver A, Lentine T, McGovern JF, Daubenspeck JA. Comparison of clinical dyspnea ratings and psychophysical measurements of respiratory sensation in obstructive airway disease. Am Rev Respir Dis. 1987 Jun;135(6):1229-33. doi: 10.1164/arrd.1987.135.6.1229. PMID 3592398
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Gencay-Can A, Can SS. Validation of the Turkish version of the fatigue severity scale in patients with fibromyalgia. Rheumatol Int. 2012 Jan;32(1):27-31. doi: 10.1007/s00296-010-1558-3. Epub 2010 Jul 24. PMID 20658235